CLINICAL TRIAL: NCT03219515
Title: Safety, Effectiveness, and Cost-effectiveness of an Herbal Medicine, Gongjin-dan, in Subjects With Chronic Dizziness: a Prospective, Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group, Clinical Trial
Brief Title: Herbal Medication (Gongjin-dan) for Chronic Dizziness
Acronym: GOODNESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyunghee University (Other)
Responsible Party: Principal Investigator, Lee Eui-ju, Professor, Ph.D. KMD., Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HB16C0010-GJD
Record Dates: First submitted 2017-07-10; First posted 2017-07-17 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Dizziness Chronic
MeSH Terms: interventions — Gongjin-dan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gongjin-dan (Experimental): Participants will be orally administered Gongjin-dan pills of 3.75g, 1 pill/day, 8 weeks (56 days).
  Interventions: Drug: Gongjin-Dan
- placebo (Placebo Comparator): Participants will be orally administered placebo pills of 3.75g, 1 pill/day, 8 weeks (56 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gongjin-Dan — Gongjin-dan (Iksu Pharmaceutical Co. Ltd, Gwangju, Republic of Korea) is composed of Cervi Parvum, Angelica Gigas Root, Cornus Fruit, Ginseng, Steamed Rehmannia Root, and Musk.
  Arms: Gongjin-dan
Drug: Placebo — Placebo drugs (similar in appearance, taste, and odor to the Gongjin-dan) contains excipients, coloring agents, binders, flavoring agents, and preservative, and gilt-paper covering. Placebo pills of Gongjin-dan will be also made by Iksu Pharmaceutical Co. Ltd, Gwangju, Republic of Korea.
  Arms: placebo

SUMMARY:
This is a prospective, multicenter, randomized, double-blinded, placebo-controlled, parallel-group, clinical trial to explore the effectiveness of an herbal medication, Gongjin-dan (GJD) for chronic dizziness (Ménière disease, psychogenic dizziness, or dizziness of unknown cause), identified as liver-deficiency pattern/syndrome, and assessed with Dizziness Handicap Inventory (DHI) ≥ 24 at baseline. Participants will be randomized and allocated to either GJD or placebo group with 1:1 ratio and orally administered GJD or placebo pills once a day for 8 weeks. For collecting data for cost-effectiveness analysis, the participants will be followed up to 12 months from randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 79 years, of either sex
2. Dizziness originating from Ménière disease, psychogenic cause, or unknown cause
3. Recurring symptom of dizziness for more than 1 month
4. Dizziness Handicap Inventory (DHI) score ≥ 24 at baseline
5. Liver-deficiency pattern/syndrome identified by Traditional Korean Medicine doctors
6. Willingness to provide written informed consent

Exclusion Criteria:

1. Dizziness attributable to vestibular disorders (e.g., benign paroxysmal positional vertigo, peripheral vestibulopathy, labyrinthitis, vestibular neuronitis, and others)
2. Dizziness attributable to central nervous system (CNS) disorders (e.g., cerebellar ataxia, stroke, demyelination, vertebrobasilar insufficiency, seizure, increased intracranial pressure, Parkinson's disease, migraines, and others)
3. Cervicogenic dizziness
4. Dizziness attributable to cardiovascular disorders (e.g., arrhythmia, heart valvular disease, anemia, orthostatic hypotension, coronary artery disease, and others)
5. Any active or uncontrolled disease that might cause dizziness (e.g., uncontrolled diabetes mellitus, hypertension, respiratory or endocrinological disorders, and others)
6. Dizziness attributable to medication side effects
7. Severe chronic or terminal diseases (malignant cancer, tuberculosis, and others)
8. Intake of other antivertiginous drugs that cannot be discontinued
9. Following physiotherapy, manual therapy (e.g., vestibular rehabilitation), and/or cognitive behavioral therapy for the treatment of dizziness
10. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen (BUN), or creatinine > 3 × upper limit of normal range at baseline
11. Women of (suspected) pregnancy or breast-feeding
12. Allergic reactions to the study medications
13. Suspicion of alcohol and/or drug abuse
14. Enrollment in another clinical study presently or within 30 days prior to the initial administration of the study medications
15. Difficulty in reliably communicating with the investigators or likelihood of inability to follow instructions
16. Other reason for ineligibility of participation

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI), change between baseline and endpoint | 56 days
  Assessment of the impairment caused by dizziness

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI), change between baseline and day 14, day 28, day 42 | 14 days
  Assessment of the impairment caused by dizziness
Mean Vertigo Score (MVS), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the intensity of dizziness
Visual Analogue Scale (VAS), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the intensity of dizziness
Frequency of episodes (dizziness), changes between baseline and day 28 and day 56 | 28 days
  The frequency score of dizziness
Berg Balance Scale (BBS), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the balance impairment
Fatigue Severity Scale (FSS), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the severity of chronic fatigue
Global Perceived Effect (GPE) | Day 56
  Assessment of a patient's perception of symptom worsening or improvement, Patient-rated outcome, 1 item, 1-7 scores
Korean version of Beck Depression Inventory (K-BDI), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the severity of depression
State-Trait Anxiety Inventory (STAI), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the severity of anxiety
Qi Blood Yin Yang deficiency questionnaire (QBYY-Q), changes between baseline and day 28 and day 56 | 28 days
  Assessment of the level of deficiency pattern/syndrome in traditional Korean medicine
EuroQol five-dimensions questionnaire five-level (EQ-5D-5L), changes between baseline and each assessment | Day 0, Day 28, Day 56, Month 4, Month 8, Month 12
  Assessment of the level of quality of life
EuroQol five dimensions questionnaire visual analogue scale (EQ VAS), change between baseline and each assessment | Day 0, Day 28, Day 56, Month 4, Month 8, Month 12
  Assessment of the level of quality of life

OTHER OUTCOMES:
Medical expenses on dizziness | Day 14, Day 28, Day 42, Day 56, Month 4, Month 8, Month 12
  medical and non-medical expenses to treat dizziness for estimating the incremental cost-effectiveness ratio
New Blinding index (New BI) | Day 56
  Blinding assessment

CONTACTS AND LOCATIONS:
Overall Officials: Euiju Lee, Ph.D., Principal Investigator — Kyunghee University
Locations (4):
- South Korea (4):
  - Dongguk University Ilsan Oriental Hospital, Goyang-si, Gyeonggi-do
  - Pusan National University Korean Medicine Hospital, Yangsan, Gyeongsangnam-do
  - Semyung University Korean Medicine Hospital, Chungju, North Chungcheong
  - Kyung Hee University Korean Medicine Hospital, Seoul, Special Seoul City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerber KA, Baloh RW. The evaluation of a patient with dizziness. Neurol Clin Pract. 2011 Dec;1(1):24-33. doi: 10.1212/CPJ.0b013e31823d07b6. PMID 23634356
- [Background] Kroenke K, Lucas CA, Rosenberg ML, Scherokman B, Herbers JE Jr, Wehrle PA, Boggi JO. Causes of persistent dizziness. A prospective study of 100 patients in ambulatory care. Ann Intern Med. 1992 Dec 1;117(11):898-904. doi: 10.7326/0003-4819-117-11-898. PMID 1443950
- [Background] Sokolova L, Hoerr R, Mishchenko T. Treatment of Vertigo: A Randomized, Double-Blind Trial Comparing Efficacy and Safety of Ginkgo biloba Extract EGb 761 and Betahistine. Int J Otolaryngol. 2014;2014:682439. doi: 10.1155/2014/682439. Epub 2014 Jun 25. PMID 25057270
- [Background] Moon E, Her Y, Lee JB, Park JH, Lee EH, Kim SH, Oh MS, Jang CG, Kim SY. The multi-herbal medicine Gongjin-dan enhances memory and learning tasks via NGF regulation. Neurosci Lett. 2009 Dec 11;466(3):114-9. doi: 10.1016/j.neulet.2009.09.033. Epub 2009 Sep 27. PMID 19788912
- [Background] Lee JS, Hong SS, Kim HG, Lee HW, Kim WY, Lee SK, Son CG. Gongjin-Dan Enhances Hippocampal Memory in a Mouse Model of Scopolamine-Induced Amnesia. PLoS One. 2016 Aug 2;11(8):e0159823. doi: 10.1371/journal.pone.0159823. eCollection 2016. PMID 27483466
- [Background] Hong SS, Lee JY, Lee JS, Lee HW, Kim HG, Lee SK, Park BK, Son CG. The traditional drug Gongjin-Dan ameliorates chronic fatigue in a forced-stress mouse exercise model. J Ethnopharmacol. 2015 Jun 20;168:268-78. doi: 10.1016/j.jep.2015.04.001. Epub 2015 Apr 10. PMID 25865680
- [Background] Sunwoo YY, Park SI, Chung YA, Lee J, Park MS, Jang KS, Maeng LS, Jang DK, Im R, Jung YJ, Park SA, Kang ES, Kim MW, Han YM. A Pilot Study for the Neuroprotective Effect of Gongjin-dan on Transient Middle Cerebral Artery Occlusion-Induced Ischemic Rat Brain. Evid Based Complement Alternat Med. 2012;2012:682720. doi: 10.1155/2012/682720. Epub 2012 Jun 6. PMID 22719787
- [Background] Son MJ, Im HJ, Kim YE, Ku B, Lee JH, Son CG. Evaluation of the anti-fatigue effects of a traditional herbal drug, Gongjin-dan, under insufficient sleep conditions: study protocol for a randomised controlled trial. Trials. 2016 Aug 22;17(1):418. doi: 10.1186/s13063-016-1542-7. PMID 27550184
- [Background] Xue Z, Liu CZ, Shi GX, Liu Y, Li ZX, Zhang ZH, Wang LP. Efficacy and safety of acupuncture for chronic dizziness: study protocol for a randomized controlled trial. Trials. 2013 Dec 13;14:429. doi: 10.1186/1745-6215-14-429. PMID 24330810
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Toupet M, Ferrary E, Grayeli AB. Visual analog scale to assess vertigo and dizziness after repositioning maneuvers for benign paroxysmal positional vertigo. J Vestib Res. 2011;21(4):235-41. doi: 10.3233/VES-2011-0420. PMID 21846956
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Hewlett S, Dures E, Almeida C. Measures of fatigue: Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF MDQ), Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales (BRAF NRS) for severity, effect, and coping, Chalder Fatigue Questionnaire (CFQ), Checklist Individual Strength (CIS20R and CIS8R), Fatigue Severity Scale (FSS), Functional Assessment Chronic Illness Therapy (Fatigue) (FACIT-F), Multi-Dimensional Assessment of Fatigue (MAF), Multi-Dimensional Fatigue Inventory (MFI), Pediatric Quality Of Life (PedsQL) Multi-Dimensional Fatigue Scale, Profile of Fatigue (ProF), Short Form 36 Vitality Subscale (SF-36 VT), and Visual Analog Scales (VAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S263-86. doi: 10.1002/acr.20579. No abstract available. PMID 22588750
- [Background] Kamper SJ, Ostelo RW, Knol DL, Maher CG, de Vet HC, Hancock MJ. Global Perceived Effect scales provided reliable assessments of health transition in people with musculoskeletal disorders, but ratings are strongly influenced by current status. J Clin Epidemiol. 2010 Jul;63(7):760-766.e1. doi: 10.1016/j.jclinepi.2009.09.009. Epub 2010 Jan 8. PMID 20056385
- [Background] Staab JP, Ruckenstein MJ. Chronic dizziness and anxiety: effect of course of illness on treatment outcome. Arch Otolaryngol Head Neck Surg. 2005 Aug;131(8):675-9. doi: 10.1001/archotol.131.8.675. PMID 16103297
- [Background] Kim J, Ku B, Kim KH. Validation of the qi blood yin yang deficiency questionnaire on chronic fatigue. Chin Med. 2016 May 2;11:24. doi: 10.1186/s13020-016-0092-y. eCollection 2016. PMID 27141228
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Derived] Shin S, Kim J, Yu A, Seo HS, Shin MR, Cho JH, Yi G, Hong SU, Lee E. A Herbal Medicine, Gongjindan, in Subjects with Chronic Dizziness (GOODNESS Study): Study Protocol for a Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Clinical Trial for Effectiveness, Safety, and Cost-Effectiveness. Evid Based Complement Alternat Med. 2017;2017:4363716. doi: 10.1155/2017/4363716. Epub 2017 Dec 13. PMID 29387128